CLINICAL TRIAL: NCT01718314
Title: Comparison of Sublingual Misoprostol Versus Lidocaine Spray for Pain Relief in Office Hysteroscopy: A Randomized, Double Blind, Placebo-Controlled Trial
Brief Title: Comparison of Sublingual Misoprostol Versus Lidocaine Spray for Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Sami Ulus Children's Hospital (Other)
Responsible Party: Principal Investigator, Sertac ESIN, Obstetrician and Gynecologist, Dr. Sami Ulus Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HEK 11/33-21
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Pain During Hysteroscopy
Keywords: Hysteroscopy; Misoprostol; Lidocaine; Visual analogue score
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sublingual Misoprostol & Lidocaine placebo (Experimental): Misoprostol 200 µg sublingually single dose and Lidocaine spray placebo
  Interventions: Drug: Sublingual Misoprostol; Drug: Placebo (for Lidocaine)
- Lidocaine Pump Spray & Misoprostol placebo (Experimental): Lidocaine Pump spray, 6 sprays to cervix (60 mg totally) and sublingual misoprotol placebo
  Interventions: Drug: Lidocaine pump spray; Drug: Placebo (for Misoprostol)

INTERVENTIONS:
Drug: Sublingual Misoprostol
  Other Names: Cytotec
  Arms: Sublingual Misoprostol & Lidocaine placebo
Drug: Lidocaine pump spray
  Other Names: Xylocaine %10 pump spray
  Arms: Lidocaine Pump Spray & Misoprostol placebo
Drug: Placebo (for Misoprostol) — Lactose filler, the pharmacy-produced pills identical to original misoprostol pill
  Arms: Lidocaine Pump Spray & Misoprostol placebo
Drug: Placebo (for Lidocaine) — The pharmacy-produced sterile saline containing pump spray external characteristics identical to lidocaine pump spray
  Arms: Sublingual Misoprostol & Lidocaine placebo

SUMMARY:
Hysteroscopy is an instrument to visualize the interior walls of uterus (womb) and it enables the doctor to do minor operative procedures. Although it causes little discomfort, sometimes it may be disturbing for the patient. This pain is usually perceived during the passage of the instrument through the cervix (neck of the womb). The investigators would like to minimize this pain by two drugs: Misoprotol and lidocaine

DETAILED DESCRIPTION:
Outpatient or office hysteroscopy has become the 'gold standard' for the investigation of the intrauterine abnormalities. This minimal invasive modality provides brilliant and clear visualization of the entire uterine cavity and besides this, by the operative channel, minor procedures may easily be performed in the office setting which is priceless for the gynecologist. However, pain related to the procedure may make the procedure uncomfortable for the patient and the physician. Together with the operative time, hysteroscope diameter is considered as the main factor influencing pain. The pain perceived during hysteroscopy may be reduced by using a smaller diameter hysteroscope or by using anesthesia, which decreases pain perception.

In this prospective, randomized, double blind, placebo controlled study, we aim to compare the effectiveness of sublingual misoprostol versus lidocaine pump spray for pain relief during office hysteroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women in the proliferative phase of the menstrual cycle with no contraindication for hysteroscopy

Exclusion Criteria:

* vaginal bleeding at the time of the procedure
* known sensitivity to lidocaine (amide group local anesthetics) or prostaglandins
* epilepsy
* significantly impaired respiratory or cardiac conduction functions
* hypertension
* glaucoma
* renal failure
* acute liver disease
* uncontrolled diabetes mellitus
* pregnancy or suspicion of pregnancy
* pelvic inflammatory disease
* cervical operation history
* vaginismus.

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Patient VAS score immediately after the procedure | Immediately after the procedure

SECONDARY OUTCOMES:
Patient VAS score 10 minutes after the procedure | 10 minutes after the procedure

OTHER OUTCOMES:
Need for cervical dilation | During the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Tuncay Kucukozkan, Professor, Study Chair — Sami Ulus Maternity and Childrens Hospital
Locations (1):
- Dr Sami Ulus Maternity and Children Training and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] van Dongen H, de Kroon CD, Jacobi CE, Trimbos JB, Jansen FW. Diagnostic hysteroscopy in abnormal uterine bleeding: a systematic review and meta-analysis. BJOG. 2007 Jun;114(6):664-75. doi: 10.1111/j.1471-0528.2007.01326.x. PMID 17516956
- [Result] De Iaco P, Marabini A, Stefanetti M, Del Vecchio C, Bovicelli L. Acceptability and pain of outpatient hysteroscopy. J Am Assoc Gynecol Laparosc. 2000 Feb;7(1):71-5. doi: 10.1016/s1074-3804(00)80012-2. PMID 10648742
- [Result] Mulayim B, Celik NY, Onalan G, Bagis T, Zeyneloglu HB. Sublingual misoprostol for cervical ripening before diagnostic hysteroscopy in premenopausal women: a randomized, double blind, placebo-controlled trial. Fertil Steril. 2010 May 1;93(7):2400-4. doi: 10.1016/j.fertnstert.2009.01.073. Epub 2009 Feb 24. PMID 19243750